CLINICAL TRIAL: NCT06609616
Title: Feasibility Of Measuring Volume of Inspiration Via Non-Invasive Motion Sensors
Brief Title: Feasibility of Measuring Volume of Inspiration Via Noninvasive Motion Sensors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10001915; 001915-CC
Record Dates: First submitted 2024-09-21; First posted 2024-09-24 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01-14

CONDITIONS: Postoperative Pulmonary Complications (PPCs)
Keywords: Measuring Volume of Inspiration; Motion Sensors; Wearable Incentive Spirometry

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Healthy participants (Experimental): Healthy participants completed a total of approximately 18 measured breaths through a traditional incentive spirometer while wearing small, non-invasive motion sensors taped to the right rib cage.
  Interventions: Device: Motion Sensor; Device: Incentive Spirometer

INTERVENTIONS:
Device: Motion Sensor — The motion sensor is the 10-axis Bluetooth Gyro Inclinometer by Wit Motion and is marketed for rehabilitation exercises, workplace injury prevention, patient care, and healthy short-range wireless motion measurements.
Device: Incentive Spirometer — A device that measures the volume of the air inhaled into the lungs during inspiration.

SUMMARY:
Background:

Lung problems develop in up to 20% of people after they have surgery. While under general anesthesia, people breathe slower and draw in less air. They may have difficulty returning to normal deep breathing as they recover. Some may develop life-threatening complications. An approved device called an incentive spirometer is used to help measure and improve a person's breathing after surgery. Researchers want to find out if a motion sensor placed on the chest can also measure the volume of air a person inhales as they breathe.

Objective:

To determine if a motion sensor on the chest can measure the volume of air a person breathes.

Eligibility:

Healthy adults aged 18 years and older.

Design:

* Participants will have one clinic visit. The visit will last 10 to 30 minutes.
* They will fill out a form with their age, sex, height, and weight.
* A small, plastic motion sensor will be taped to their chest on one or both sides.
* Participants will breathe through a tube attached to an incentive spirometer. They will take 18 breaths of different volumes, both deep and shallow.
* Researchers will use the data collected from the motion sensors to measure how the chest moves at different levels of breathing. The motion sensor data will be used to create a software program that converts chest wall motion to the volume of air inhaled for a given breath in real time.

DETAILED DESCRIPTION:
Study Description:

This protocol is a basic physiologic proof-of-concept study enrolling normal volunteers to determine the feasibility of measuring volume of inspiration from chest wall motion measured via non-invasive thoracic motion sensors. The motion sensors are not medical devices because they are not intended to diagnose a disease or condition or to cure, mitigate, treat or prevent disease. Since motion sensors are not being evaluated for diagnostic purposes or being studied themselves within the context of this protocol and are only intended to collect physiological data, they are not to be considered investigational. The data collected in this feasibility study will not contain any personally identifiable information (PII). In this study, healthy participants will complete a total of approximately 18 measured breaths through a traditional incentive spirometer while wearing small, non-invasive motion sensors on their thorax at approximately the level of the 9th and 10th ribs unilaterally or bilaterally. The incentive spirometer is an FDA approved medical device. This study does not aim to study the safety or effectiveness of this device but rather utilize the device as a tool to measure volume of inspiration. The waveform data collected from the devices with each breath will then be analyzed with the intention to develop an algorithm that could convert chest wall motion to a discrete volume of inspiration in real time. Total enrollment time will be about 10-30 minutes per participant.

Objectives:

Primary: To collect chest wall motion data corresponding to various volumes of inspiration from a non-invasive wearable device.

Secondary: To develop an algorithm which can convert chest wall motion to volume of inspiration and assess the algorithm using cross-validation strategy.

Endpoints:

Primary: A database of motion waveforms corresponding to each measured volume of inspiration via traditional incentive spirometer.

Secondary: A cross-validated algorithm that converts chest wall motion to volume of inspiration.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this proof-of-concept study, an individual must meet all the following criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female sex, aged 18-100.
4. Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Pregnancy.
2. Known allergic reactions to adhesive.
3. Patients with an altered mental status that precludes understanding and consenting for the procedure and compliance with the study activities.
4. Patients with known pulmonary conditions including pulmonary fibrosis, asthma, chronic obstructive pulmonary disease (COPD), or chronic bronchitis.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Pinto, M.D., Principal Investigator — National Institutes of Health, National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing complies with the institution's data management and sharing (DMS) policy
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From study completion
Access Criteria: This study complies with the National Institutes of Health (NIH) public access policy, which ensures that the public has access to the published results of NIH funded research.
  Data can also be provided to investigators for future study upon written request.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001915-CC.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Participants
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Participants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 7
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Secondary Outcome: Participants With Convertible Chest Wall Motion Waveform
Description: Participants with waveform data that support the development and and validation of an algorithm that converts chest-wall motion waveforms into estimated volumes of inspiration. For each participant, motion waveforms is annotated with the corresponding measured inspiratory volumes.
Time Frame: Within a month of study completion
Population: The analyses included all participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants
Number analyzed (Participants) | 30
Participants | 30

2. Primary Outcome: Participants With Collectable Waveform Data
Description: Number of participants with collectable waveform data, which corresponds to each breathing exercise from the wearable motion sensor and uploaded to a secured database.
Time Frame: 15-20 minutes from start of the study
Population: The analyses included all participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants
Number analyzed (Participants) | 30
Participants | 30

ADVERSE EVENTS:
Time Frame: 15-30 minutes within procedure and 30 minutes after procedure, for a maximum of one hour
Arm/Group | Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT06609616/Prot_SAP_000.pdf